CLINICAL TRIAL: NCT03201120
Title: Reducing UV Exposure to Prevent Skin Cancer: Message Development & Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Glanz, Professor of Epidemiology and Nursing, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 821348
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor Sun Exposure Behavior (Experimental): A convenience sample of white, English-speaking adults ages 18 to 49 will be recruited via online advertisements in Philadelphia and the surrounding region (within a 30 mile radius). The investigators will recruit 120 adults to test outdoor UV exposure messages. The investigators will quota sample to ensure representation across age and gender groups.
  The inclusion criteria are that adults must be white, must be between 18-49 years old and must speak English.
  Interventions: Behavioral: Outdoor Sun Behavior
- Indoor Tanning Behavior (Experimental): A convenience sample of white, English-speaking females ages 18 to 25 will be recruited via online advertisements and flyers in Philadelphia and the surrounding region (within a 30 mile radius). The investigators will recruit 60 adults to test indoor tanning messages.
  The inclusion criteria are that adults must be white, female, must be between 18-25 years old, must have used an indoor tanning bed at least once in the past 12 months, and must speak English.
  Interventions: Behavioral: Indoor Tanning Behavior

INTERVENTIONS:
Behavioral: Outdoor Sun Behavior — Participants will provide informed consent and complete a short background questionnaire about usual sun exposure and protection behaviors and demographics. Next, each participant will be seated in a room to view the audio-visual media messages. Eye-tracking equipment running Paradigm (Perception Research Systems Incorporated) for stimuli presentation will be calibrated to the participant. Subjects will be seated at a desk in front of a computer monitor, keyboard and mouse setup. Each participant will view messages with different emotional appeals related to outdoor sun exposure (seeking shade, covering up, using sunscreen, and multiple behaviors). Messages will be shown in random order, with each message interspersed by a 30 second baseline screen consisting of black background and white, centered plus sign. The last 10 seconds of each preceding the 30-second baseline screen will be used to establish physiologic baseline to minimize carry-over effects of the preceding message.
  Arms: Outdoor Sun Exposure Behavior
Behavioral: Indoor Tanning Behavior — Upon arrival, participants will provide informed consent and complete a short background questionnaire about usual indoor tanning, sun exposure and protection behaviors, and demographics. Next, each participant will be seated in a room to view the audio-visual media messages. Eye-tracking equipment running Paradigm (Perception Research Systems Incorporated) for stimuli presentation will be calibrated to the participant. Subjects will be seated at a desk in front of a typical computer monitor, keyboard and mouse setup. Each participant will view messages with each type of target behavior (freedom, health risk, appearance)). Messages will be shown in random order, with each message interspersed by a 30 second baseline screen consisting of black background and white, centered plus sign. The last 10 seconds of each preceding the 30-second baseline screen will be used to establish physiologic baseline to minimize carry-over effects of the preceding message.
  Arms: Indoor Tanning Behavior

SUMMARY:
Phase 3b of the research will be a laboratory experiment that uses an experimental and analytic design that is parallel to that used in Phase 3a, the online experiment. The primary objective of Phase 3b is to assess physiological response (i.e., eye tracking) to different message appeals of the audio-visual messages used in Phase 3a on respondents' behavioral intentions and UV-related behavioral choices post-exposure. Including time for preparation, viewing, and removal of the monitoring equipment, the message viewing session will take about 45 minutes per session.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 year old non-Hispanic white (NHW) adults
* OR 18-25 year old NHW females who have tanned indoors in the past 12 months

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3595 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Laboratory Survey | Baseline
  Questionnaire measures will be completed using an iPad with Qualtrics software. Participants will be asked to evaluate each message for its argument strength, emotional appeal, and themes; participants will also be asked about their intentions and beliefs related to each behavior. The research technician will not initiate a conversation with the participant during the experimental session except to give instructions.
Follow-up Survey | Two weeks post baseline Laboratory Survey
  Two weeks after the completed laboratory session, participants will be emailed a link to complete a follow-up survey. The survey will ask about participants' ability to recall the messages, attitudes regarding outdoor sun protection behaviors, actual behaviors in the past two weeks, whether the participants have used or will use the product they selected, and whether the participants have discussed the messages with anyone else.

SECONDARY OUTCOMES:
Measure of Behavioral Intent | Baseline
  Upon finishing the experiment, respondents will be offered a choice of one of four "thank you" gifts of comparable value: sunscreen, hand sanitizer, and moisturizer with or without SPF protection. The experimenter will unobtrusively record the subjects' selections.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- CIRNA Lab, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No